CLINICAL TRIAL: NCT00645801
Title: Lubiprostone Plus Polyethylene Glycol-electrolyte Solutionvs. Placebo Plus Polyethylene Glycol-electrolyte Solution for Outpatient Colonoscopy Preparation: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Amitiza® Plus GoLYTELY® (PEG) Versus Placebo Plus GoLYTELY® for Outpatient Colonoscopy Preparation
Acronym: PEG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Ann L. Silverman, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-024L
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Results first posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Colonoscopy
Keywords: Routine screening colonoscopy; Colonoscopy Preparation; Amitiza; GoLYTELY; Pegylated Electrolytes; Preparation Solution; Colonoscopy Solution
MeSH Terms: interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinding was done to ensure minimum bias. The clinicians attending to the patients were not involved in the randomization process, and all were blinded to the identity of the drug received as the placebo was identical to the active drug in packaging, appearance, and schedule of administration. Separate individuals generated the allocation sequence, enrolled participants, and assigned participants to their groups. The blind was maintained until all decisions regarding data evaluability were made. Only the research assistant who assigned participants to their treatment groups was permitted access to the randomization list, which was maintained in a locked filing cabinet during the trial. The patients were blinded to their medication status.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ingested 4 tablets of lubiprostone in divided doses + 1 gallon of polyethylene glycol (Active Comparator): First dose of lubiprostone 24 micrograms or placebo was administered 2 nights before colonoscopy and subsequent doses at breakfast, lunch, and dinner on the day before the procedure. Patients were on a clear liquid diet on the day before the procedure and were instructed to initiate drinking PEG (immediately after the last dose of lubiprostone) at 6 PM the evening before the colonoscopy and continued drinking the solution until at least 2 bowel movements were clear yellow or green. All study patients were educated and instructed to observe for clear stool, which was defined as "watery consistency without any solid fecal material or dark liquid stools." Patients were instructed to return the unused PEG solution on the day of colonoscopy. After completing the preparation but before colonoscopy, patients were also required to fill a questionnaire to assess the tolerability of tablets and solution.
  Interventions: Drug: lubiprostone (Amitiza)
- Ingested 4 tablets of placebo in divided doses + 1 gallon of polyethylene glycol (Placebo Comparator): First dose of look alike placebo was administered 2 nights before colonoscopy and subsequent doses at breakfast, lunch, and dinner on the day before the procedure. Patients were on a clear liquid diet on the day before the procedure and were instructed to initiate drinking PEG (immediately after the last dose of lubiprostone) at 6 PM the evening before the colonoscopy and continued drinking the solution until at least 2 bowel movements were clear yellow or green. All study patients were educated and instructed to observe for clear stool, which was defined as "watery consistency without any solid fecal material or dark liquid stools." Patients were instructed to return the unused PEG solution on the day of colonoscopy. After completing the preparation but before colonoscopy, patients were also required to fill a questionnaire to assess the tolerability of tablets and solution.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lubiprostone (Amitiza) — 24 mcg administered 4 times over the two days before the colonoscopy. 96 mcg total
  Other Names: Amitiza
  Arms: Ingested 4 tablets of lubiprostone in divided doses + 1 gallon of polyethylene glycol
Drug: Placebo — Amitiza Placebo
  Other Names: Look alike placebo Amitiza
  Arms: Ingested 4 tablets of placebo in divided doses + 1 gallon of polyethylene glycol

SUMMARY:
The primary objective is to compare the effectiveness and tolerance of the medication named lubiprostone plus a large volume liquid laxative versus placebo which is a look alike medication that has no effect such as a sugar pill plus a large volume liquid laxative as a bowel cleaning preparation for colonoscopy to see the colon better during the colonoscopy to identify abnormal growths such as polyps or colon cancer.

Colonoscopy is considered the best way to screen for colon cancer screening because you can visualize the colon directly and remove or biopsy abnormal growths. The limiting step in the procedure is the quality of the colon preparation prior to the procedure. Many patients do not tolerate large volumes of liquid used to prepare the colon. The purpose of the study is to improve the quality of the prep by adding a pill laxative medication before starting the large volume laxative to better see the colon. The other aim of the study is to try to reduce the amount of of liquid laxative the patient has to drink by giving a pill laxative before starting the liquid laxative.

DETAILED DESCRIPTION:
The study is a double blind placebo controlled study of lubiprostone in 4 doses vs look alike placebo in 4 doses before bowel preparation for outpatient screening, surveillance and diagnostic colonoscopy. Patients with severe underlying medical conditions were excluded. Patients with inflammatory bowel disease, frequent bowel movements and colonic resection were also excluded. Patients were randomized to one of two groups. The study was double blinded. The first group took lubiprostone 24 micrograms and the second group took look alike placebo in 4 divided doses right before starting the bowel prep with the last dose upon starting polyethylene glycol-electrolyte solution the evening before the colonoscopy.

All study patients were educated and instructed to observe for clear stool, which was defined as "watery consistency without any solid fecal material or dark liquid stools" before stopping the liquid bowel prep. Patients were instructed to return the unused PEG solution on the day of colonoscopy. After completing the preparation but before colonoscopy, patients were also required to fill a questionnaire to assess the tolerability of tablets and solution. This was measured on a 1-5 rating Likert scale (1) "Easy," 2) "Tolerable," 3) "Slightly Difficult," 4) "Extremely Difficult," and 5)"Unable to Finish" and was based on the patient's ability to swallow the liquid and each of 4 tablets. In addition, the pres- ence of symptoms of nausea, vomiting, abdominal pain, chest pain, dizziness, and bloating was evaluated.

The primary endpoints was the endoscopist's evaluation of the preparation quality. All colonoscopies were performed by 3 endoscopists (with 85% of the procedures performed by principal investigator of the study, A.L.S.). Endo- scopists evaluated the quality of the colonoscopy prep- aration based on the previously validated Ottawa bowel preparation scale.5 This scale rates 3 sections of colon, rectosigmoid, mid, and right colon, on a 5-point scale (0-4) and a global 3-point rating (0-2) for overall colonic fluid. The total score ranges from 0-14; score of 0 being perfect and score of 14 indicating solid stool in each colon segment and lot of fluid.The secondary endpoint was to determine any reduction in the amount of PEG consumed in the lubiprostone group compared with the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years old
* Subject is in good health
* Subject is undergoing a screening, surveillance or diagnostic colonoscopy
* Subject has a spontaneous bowel movement at least every 48 hours

Exclusion Criteria:

* Subject has renal insufficiency demonstrated by serum creatinine > 1.4mg/dL
* Subject has Type 1 diabetes
* Subject has past or present diagnosis of Congestive Heart Failure
* Subject has past or present diagnosis of inflammatory bowel disease
* Subject had previous colon resection
* Subject has a preexisting electrolyte abnormality
* Subject has more than 3 spontaneous bowel movements daily

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2008-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann L Silverman, MD, Principal Investigator — Henry Ford Health System
Locations (3):
- United States (3):
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health System, Novi, Michigan
  - Henry Ford Health System, West Bloomfield, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Froehlich F, Wietlisbach V, Gonvers JJ, Burnand B, Vader JP. Impact of colonic cleansing on quality and diagnostic yield of colonoscopy: the European Panel of Appropriateness of Gastrointestinal Endoscopy European multicenter study. Gastrointest Endosc. 2005 Mar;61(3):378-84. doi: 10.1016/s0016-5107(04)02776-2. PMID 15758907
- [Background] Harewood GC, Sharma VK, de Garmo P. Impact of colonoscopy preparation quality on detection of suspected colonic neoplasia. Gastrointest Endosc. 2003 Jul;58(1):76-9. doi: 10.1067/mge.2003.294. PMID 12838225
- [Background] Afridi SA, Barthel JS, King PD, Pineda JJ, Marshall JB. Prospective, randomized trial comparing a new sodium phosphate-bisacodyl regimen with conventional PEG-ES lavage for outpatient colonoscopy preparation. Gastrointest Endosc. 1995 May;41(5):485-9. doi: 10.1016/s0016-5107(05)80008-2. PMID 7615228
- [Background] Johanson JF, Ueno R. Lubiprostone, a locally acting chloride channel activator, in adult patients with chronic constipation: a double-blind, placebo-controlled, dose-ranging study to evaluate efficacy and safety. Aliment Pharmacol Ther. 2007 Jun 1;25(11):1351-61. doi: 10.1111/j.1365-2036.2007.03320.x. PMID 17509103
- [Background] Camilleri M, Bharucha AE, Ueno R, Burton D, Thomforde GM, Baxter K, McKinzie S, Zinsmeister AR. Effect of a selective chloride channel activator, lubiprostone, on gastrointestinal transit, gastric sensory, and motor functions in healthy volunteers. Am J Physiol Gastrointest Liver Physiol. 2006 May;290(5):G942-7. doi: 10.1152/ajpgi.00264.2005. PMID 16603730
- [Background] Stengel JZ, Jones DP. Single-dose lubiprostone along with split-dose PEG solution without dietary restrictions for bowel cleansing prior to colonoscopy: a randomized, double-blind, placebo-controlled trial. Am J Gastroenterol. 2008 Sep;103(9):2224-30. doi: 10.1111/j.1572-0241.2008.02053.x. Epub 2008 Aug 5. PMID 18684185
- [Background] Grigg E, Schubert MC, Hall J, Rahhal F, Raina D, Sridhar S, Chamberlain SM. Lubiprostone used with polyethylene glycol in diabetic patients enhances colonoscopy preparation quality. World J Gastrointest Endosc. 2010 Jul 16;2(7):263-7. doi: 10.4253/wjge.v2.i7.263. PMID 21160617
- [Background] Park JS, Sohn CI, Hwang SJ, Choi HS, Park JH, Kim HJ, Park DI, Cho YK, Jeon WK, Kim BI. Quality and effect of single dose versus split dose of polyethylene glycol bowel preparation for early-morning colonoscopy. Endoscopy. 2007 Jul;39(7):616-9. doi: 10.1055/s-2007-966434. PMID 17611916
- [Background] Aoun E, Abdul-Baki H, Azar C, Mourad F, Barada K, Berro Z, Tarchichi M, Sharara AI. A randomized single-blind trial of split-dose PEG-electrolyte solution without dietary restriction compared with whole dose PEG-electrolyte solution with dietary restriction for colonoscopy preparation. Gastrointest Endosc. 2005 Aug;62(2):213-8. doi: 10.1016/s0016-5107(05)00371-8. PMID 16046981
- [Background] Marmo R, Rotondano G, Riccio G, Marone A, Bianco MA, Stroppa I, Caruso A, Pandolfo N, Sansone S, Gregorio E, D'Alvano G, Procaccio N, Capo P, Marmo C, Cipolletta L. Effective bowel cleansing before colonoscopy: a randomized study of split-dosage versus non-split dosage regimens of high-volume versus low-volume polyethylene glycol solutions. Gastrointest Endosc. 2010 Aug;72(2):313-20. doi: 10.1016/j.gie.2010.02.048. Epub 2010 Jun 19. PMID 20561621
- [Background] Unger RZ, Amstutz SP, Seo DH, Huffman M, Rex DK. Willingness to undergo split-dose bowel preparation for colonoscopy and compliance with split-dose instructions. Dig Dis Sci. 2010 Jul;55(7):2030-4. doi: 10.1007/s10620-009-1092-x. Epub 2010 Jan 16. PMID 20082216
- [Background] American Society of Anesthesiologists Committee. Practice guidelines for preoperative fasting and the use of pharmacologic agents to reduce the risk of pulmonary aspiration: application to healthy patients undergoing elective procedures: an updated report by the American Society of Anesthesiologists Committee on Standards and Practice Parameters. Anesthesiology. 2011 Mar;114(3):495-511. doi: 10.1097/ALN.0b013e3181fcbfd9. No abstract available. PMID 21307770
- [Background] Park SS, Sinn DH, Kim YH, Lim YJ, Sun Y, Lee JH, Kim JY, Chang DK, Son HJ, Rhee PL, Rhee JC, Kim JJ. Efficacy and tolerability of split-dose magnesium citrate: low-volume (2 liters) polyethylene glycol vs. single- or split-dose polyethylene glycol bowel preparation for morning colonoscopy. Am J Gastroenterol. 2010 Jun;105(6):1319-26. doi: 10.1038/ajg.2010.79. Epub 2010 May 18. PMID 20485282
- [Background] Abdul-Baki H, Hashash JG, Elhajj II, Azar C, El Zahabi L, Mourad FH, Barada KA, Sharara AI. A randomized, controlled, double-blind trial of the adjunct use of tegaserod in whole-dose or split-dose polyethylene glycol electrolyte solution for colonoscopy preparation. Gastrointest Endosc. 2008 Aug;68(2):294-300; quiz 334, 336. doi: 10.1016/j.gie.2008.01.044. Epub 2008 Jun 3. PMID 18511049
- [Background] Hookey LC, Depew WT, Vanner SJ. Combined low volume polyethylene glycol solution plus stimulant laxatives versus standard volume polyethylene glycol solution: a prospective, randomized study of colon cleansing before colonoscopy. Can J Gastroenterol. 2006 Feb;20(2):101-5. doi: 10.1155/2006/621367. PMID 16482236
- [Background] Taylor C, Schubert ML. Decreased efficacy of polyethylene glycol lavage solution (golytely) in the preparation of diabetic patients for outpatient colonoscopy: a prospective and blinded study. Am J Gastroenterol. 2001 Mar;96(3):710-4. doi: 10.1111/j.1572-0241.2001.03610.x. PMID 11280539
- [Background] Siddiqui AA, Yang K, Spechler SJ, Cryer B, Davila R, Cipher D, Harford WV. Duration of the interval between the completion of bowel preparation and the start of colonoscopy predicts bowel-preparation quality. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):700-6. doi: 10.1016/j.gie.2008.09.047. PMID 19251013
- [Background] Rostom A, Jolicoeur E. Validation of a new scale for the assessment of bowel preparation quality. Gastrointest Endosc. 2004 Apr;59(4):482-6. doi: 10.1016/s0016-5107(03)02875-x. PMID 15044882

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two hundred patients were planned to enroll in the study; however, the study was discontinued by the sponsor before the enrollment goal was completed because of slow enrollment. Of the 157 patients who volunteered for the study, only 123 patients who actually did the bowel preparation. Patients were recruited from the gastroenterology clinic at the main hospital and at the satellite clinic in the suburbs of Detroit.
Pre-assignment Details: Exclusion criteria included serum creatinine greater than 1.4, type I diabetes, CHF, pre-existing electrolyte abnormalities, inflammatory bowel disease, no spontaneous bowel movement every 48 hours, more than 3 bowel movements daily and previous colon resection.
Groups:
- 1 Patient Received Both Lubiprostone in 4 Divided Doses and Golytely.: First dose of lubiprostone was administered 2 nights before colonoscopy and subsequent doses at breakfast, lunch, and dinner on the day before the procedure. Patients were instructed to initiate drinking PEG (immediately after the last dose of lubiprostone) at 6 PM the evening before the colonoscopy and continued drinking the solution until at least 2 bowel movements were clear yellow or green. After completing the preparation but before colonoscopy, patients were also required to fill a questionnaire to assess the tolerability of tablets and solution. This was measured on a 1-5 rating Likert scale 1) Easy, up to 5) Unable to Finish. In addition, the presence of symptoms of nausea, vomiting, abdominal pain, chest pain, dizziness, and bloating was also noted. All colonoscopies were performed by 3 endoscopists (with 85% of the procedures performed by principal investigator of the study, A.L.S.). Endoscopists evaluated the quality of the colonoscopy preparation based on the Ottawa bowel preparation scale. This scale rates 3 sections of colon, rectosigmoid, mid, and right colon, on a 5-point scale (0-4) and a global 3-point rating (0-2) for overall colonic fluid. The total score ranges from 0-14; score of 0 being perfect and score of 14 indicating solid stool in each colon segment and lot of fluid. All patients were contacted by telephone the day after the procedure to determine if they were experiencing any adverse reactions.
- 2 Look Alike Placebo in 4 Divided Doses Plus PEG and Electrolytes.: group 2 ingested 4 tablets of placebo (in divided doses) + 1 gallon of PEG. First dose of placebo was administered 2 nights before colonoscopy and subsequent doses at breakfast, lunch, and dinner on the day before the procedure. Patients were instructed to initiate drinking PEG (immediately after the last dose of lubiprostone) at 6 PM the evening before the colonoscopy and continue drinking the solution until at least 2 bowel movements were clear yellow or green. Patients evaluated the prep on a 1-5 rating Likert scale 1)Easy, to 5) Unable to Finish In addition, the presence of symptoms of nausea, vomiting, abdominal pain, chest pain, dizziness, and bloating were also recorded.All colonoscopies were performed by 3 endoscopists (with 85% of the procedures performed by principal investigator of the study, A.L.S.). Endoscopists evaluated the quality of the colonoscopy preparation based on the Ottawa bowel preparation scale. This scale rates 3 sections of colon, rectosigmoid, mid, and right colon, on a 5-point scale (0-4) and a global 3-point rating (0-2) for overall colonic fluid. The total score ranges from 0-14; score of 0 being perfect and score of 14 indicating solid stool in each colon segment and lot of fluid. All patients were contacted by telephone the day after the procedure to determine if they were experiencing any adverse reactions.
Period: Overall Study
Arm/Group | 1 Patient Received Both Lubiprostone in 4 Divided Doses and Golytely. | 2 Look Alike Placebo in 4 Divided Doses Plus PEG and Electrolytes.
Started | 77 | 81
Completed | 57 | 66
Not Completed | 20 | 15
Not completed — unclear if patient took all the medication. | 1 | 0
Not completed — Lost to Follow-up | 19 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 Look Alike Placebo in 4 Divided Doses Plus PEG and Electrolytes. | 1 Patient Received Both Lubiprostone in 4 Divided Doses and Golytely. | Total
Number analyzed (Participants) | 66 | 57 | 123
Age, Continuous [Mean (Standard Deviation); unit: years]
  age | 56.1 (9.1) | 55.8 (9.4) | 56.0 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 35 | 76
  Male | 25 | 22 | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 66 | 57 | 123

OUTCOME MEASURES:

1. Primary Outcome: Endoscopist Evaluation of Colon Cleanliness in the Lubiprostone Group vs the Placebo Group
Description: Endoscopists evaluated the quality of the colonoscopy preparation based on Ottawa bowel preparation scale. . The total score ranges from 0-14; score of 0 being perfect and score of 14 indicating solid stool in each colon segment and lot of fluid. Before using the scale for this trial, the endoscopists participated in a calibration exercise that involved 20 patients to ensure that they concurred on their interpretation of the scale.
Time Frame: within 12 hours of completing bowel prep
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Look Alike Placebo in 4 Divided Doses Plus PEG and Electrolytes.: group 2 ingested 4 tablets of placebo (in divided doses) + 1 gallon of PEG. First dose of placebo was administered 2 nights before colonoscopy and subsequent doses at breakfast, lunch, and dinner on the day before the procedure. Patients were instructed to initiate drinking PEG (immediately after the last dose of lubiprostone) at 6 PM the evening before the colonoscopy and continue drinking the solution until at least 2 bowel movements were clear yellow or green. Patients evaluated the prep on a 1-5 rating Likert scale 1)Easy, to 5) Unable to Finish In addition, the presence of symptoms of nausea, vomiting, abdominal pain, chest pain, dizziness, and bloating were also recorded.All colonoscopies were performed by 3 endoscopists (with 85% of the procedures performed by principal investigator of the study, A.L.S.). Endoscopists evaluated the quality of the colonoscopy preparation based on the Ottawa bowel preparation scale. This scale rates 3 sections of colon, rectosigmoid, mid, and right colon, on a 5-point scale (0-4) and a global 3-point rating (0-2) for overall colonic fluid. The total score ranges from 0-14; score of 0 being perfect and score of 14 indicating solid stool in each colon segment and lot of fluid. All patients were contacted by telephone the day after the procedure to determine if they were experiencing any adverse reactions.
- Patient Received Both Lubiprostone in 4 Divided Doses and Golytely.: First dose of lubiprostone was administered 2 nights before colonoscopy and subsequent doses at breakfast, lunch, and dinner on the day before the procedure. Patients were instructed to initiate drinking PEG (immediately after the last dose of lubiprostone) at 6 PM the evening before the colonoscopy and continued drinking the solution until at least 2 bowel movements were clear yellow or green. After completing the preparation but before colonoscopy, patients were also required to fill a questionnaire to assess the tolerability of tablets and solution. This was measured on a 1-5 rating Likert scale 1) Easy, up to 5) Unable to Finish. In addition, the presence of symptoms of nausea, vomiting, abdominal pain, chest pain, dizziness, and bloating was also noted. All colonoscopies were performed by 3 endoscopists (with 85% of the procedures performed by principal investigator of the study, A.L.S.). Endoscopists evaluated the quality of the colonoscopy preparation based on the Ottawa bowel preparation scale. This scale rates 3 sections of colon, rectosigmoid, mid, and right colon, on a 5-point scale (0-4) and a global 3-point rating (0-2) for overall colonic fluid. The total score ranges from 0-14; score of 0 being perfect and score of 14 indicating solid stool in each colon segment and lot of fluid. All patients were contacted by telephone the day after the procedure to determine if they were experiencing any adverse reactions.
Arm/Group | Look Alike Placebo in 4 Divided Doses Plus PEG and Electrolytes. | Patient Received Both Lubiprostone in 4 Divided Doses and Golytely.
Number analyzed (Participants) | 66 | 57
score on a scale | 1.38 (0.49) | 1.24 (0.59)
Statistical Analysis 1: Comparison: Look Alike Placebo in 4 Divided Doses Plus PEG and Electrolytes. vs Patient Received Both Lubiprostone in 4 Divided Doses and Golytely; Based on the assumption that 70% of patients using PEG plus placebo (group 2) will have good results, by allocating 100 cases in each group, we will have 84% power to detect a difference of 18% or more in the effectiveness of PEG plus lubiprostone combination (group 1) (eg, 70% in group 2 vs. 88% in group 1) at the alpha level of significancelevel of significance; Test type: Superiority; p = 0.05, t-test, 2 sided — A 2-sided 2 sample t test was used to compare the overall cleanliness score between the 2 treatment groups

2. Secondary Outcome: Tolerability of the Colon Cleansing Group in the Lubiprostone Group vs the Placebo Group
Description: After completing the colonoscopy prep patients were asked to assess tolerability of the prep using a 5 point Likert scale with 1 being easy and 5 being unable to complete the prep
Time Frame: done at the time of colonoscopy
Population: Patients completed the drug or placebo with PEG and completed a questionnaire on the day of of the colonoscopy
Measure: Number; unit: participants
Groups:
- Ingested 4 Tablets of Lubiprostone in Divided Doses + 1 Gallon of Polyethylene Glycol: First dose of lubiprostone 24 micrograms or placebo was administered 2 nights before colonoscopy and subsequent doses at breakfast, lunch, and dinner on the day before the procedure. before colonoscopy, patients were also required to fill a questionnaire to assess the tolerability of tablets and solution. Patient tolerability was determined on a 5 point likert scale after completing the prep.
  lubiprostone (Amitiza): 24 mcg administered 4 times over the two days before the colonoscopy. 96 mcg total
- Ingested 4 Tablets of Placebo in Divided Doses + 1 Gallon of Polyethylene Glycol: First dose of look alike placebo was administered 2 nights before colonoscopy and subsequent doses at breakfast, lunch, and dinner on the day before the procedure. Patient tolerability was determined on a 5 point Likert scale.
  Placebo: Amitiza Placebo
Arm/Group | Ingested 4 Tablets of Lubiprostone in Divided Doses + 1 Gallon of Polyethylene Glycol | Ingested 4 Tablets of Placebo in Divided Doses + 1 Gallon of Polyethylene Glycol
Number analyzed (Participants) | 52 | 64
participants
  easy | 6 | 4
  Tolerable | 15 | 14
  slightly difficult | 18 | 25
  extremely difficult | 6 | 15
  unable to finish | 7 | 6
Statistical Analysis 1: Comparison: Ingested 4 Tablets of Lubiprostone in Divided Doses + 1 Gallon of Polyethylene Glycol vs Ingested 4 Tablets of Placebo in Divided Doses + 1 Gallon of Polyethylene Glycol; Test type: Superiority; p < 0.05, 2 sided Cochran-Armitage trend test

3. Secondary Outcome: Change in Volume of PEG From Beginning of Bowel Prep to That at Completion of the Colonoscopy Preparation in the Two Groups
Description: Patients in the lubiprostone group and the placebo returned unused PEG after completing the prep for the colonoscopy. This was measured in liters and recorded.
Time Frame: amount of PEG at start of the study and that measured when the patient presented for their procedure.
Measure: Mean (Standard Deviation); unit: liters
Groups:
- Ingested 4 Tablets of Placebo in Divided Doses + 1 Gallon of Polyethylene Glycol: First dose of look alike placebo was administered 2 nights before colonoscopy and subsequent doses at breakfast, lunch, and dinner on the day before the procedure. n.
  Placebo: Amitiza Placebo
- Ingested 4 Tablets of Lubiprostone in Divided Doses + 1 Gallon of Polyethylene Glycol: First dose of lubiprostone 24 micrograms or placebo was administered 2 nights before colonoscopy and subsequent doses at breakfast, lunch, and dinner on the day before the procedure. .
  lubiprostone (Amitiza): 24 mcg administered 4 times over the two days before the colonoscopy. 96 mcg total
Arm/Group | Ingested 4 Tablets of Placebo in Divided Doses + 1 Gallon of Polyethylene Glycol | Ingested 4 Tablets of Lubiprostone in Divided Doses + 1 Gallon of Polyethylene Glycol
Number analyzed (Participants) | 57 | 66
liters | 0.79 (0.97) | 1.36 (1.04)
Statistical Analysis 1: Comparison: Ingested 4 Tablets of Placebo in Divided Doses + 1 Gallon of Polyethylene Glycol vs Ingested 4 Tablets of Lubiprostone in Divided Doses + 1 Gallon of Polyethylene Glycol; Test type: Superiority; p < 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 2 days that the patients took lubiprostone or placebo.
Description: Patients were asked to describe any symptoms during colonoscopy prep
Groups:
- Ingested 4 Tablets of Lubiprostone in Divided Doses + 1 Gallon of Polyethylene Glycol: lubiprostone (Amitiza): 24 mcg administered 4 times over the two days of the colon preparation with PEG plus electrolytes before the colonoscopy. 96 mcg total lubiprostone
- Ingested 4 Tablets of Placebo in Divided Doses + 1 Gallon of Polyethylene Glycol: Placebo: Amitiza Placebo 4 times over the two days of the colon preparation in divided doses with PEG plus electrolytes before the colonoscopy.
Arm/Group | Ingested 4 Tablets of Lubiprostone in Divided Doses + 1 Gallon of Polyethylene Glycol | Ingested 4 Tablets of Placebo in Divided Doses + 1 Gallon of Polyethylene Glycol
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/66
Other Adverse Events (participants affected / at risk) | 41/57 | 46/66
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ingested 4 Tablets of Lubiprostone in Divided Doses + 1 Gallon of Polyethylene Glycol (N=57) | Ingested 4 Tablets of Placebo in Divided Doses + 1 Gallon of Polyethylene Glycol (N=66)
nausea (Gastrointestinal disorders) | 21 | 25
bloating (Gastrointestinal disorders) | 9 | 13
headache (Nervous system disorders) | 6 | 3
abdominal pain (Gastrointestinal disorders) | 0 | 3
flatulence (Gastrointestinal disorders) | 0 | 2
Tingling of extremities (Nervous system disorders) | 1 | 1
anal irritation (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No